CLINICAL TRIAL: NCT05920330
Title: Novel Mechanisms and Therapeutic Approaches for Nasal Obstruction and Olfactory Losses
Brief Title: Nasal Obstruction and Olfactory Losses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kai Zhao, Associate Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015H0262
Record Dates: First submitted 2023-05-22; First posted 2023-06-27 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Nasal Obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Intervention Model Description: Patients experiencing olfactory impairment and/or nasal obstruction, self-referred to participate in the research study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): A device-nasal plug will be self-inserted into the nose with a diagonal channel embedded to redirect nasal airflow patterns to different nasal regions. A nose clip will be used to pinch the nose externally, similar to what synchronized swimmers use.
  Interventions: Other: Nasal Plug

INTERVENTIONS:
Other: Nasal Plug — Please see the arm description for details.
  Other Names: Swimmer's nose clip

SUMMARY:
About 13% of US adults, some 30 million people, suffer from nasal sinus disease. Although nasal obstruction and smell loss are two of the major symptoms of the disease that are crucial to disease management, currently there is a lack of clinical tools to effectively evaluate the mechanisms contributing to these symptoms. The proposed study aims to develop novel clinical tools to better evaluate and relieve patients' nasal obstructive symptoms and to enable patients and clinicians to make more informed, personalized decisions regarding treatment strategy.

DETAILED DESCRIPTION:
Nasal sinus disease is one of the most common medical conditions in the US, affecting an estimated 13% of adults, or some 30 million people, and responsible for $5.8 billion in health care expenditures annually (National Health Interview Survey 2009, CDC). Nasal obstruction and smell loss are two of the major symptoms of the disease; however, the field currently lacks a clear, objective understanding of the mechanisms causing these symptoms, which thwarts effective treatment. For example, patients' complaints of nasal obstruction correlate poorly or inconsistently with objective measurements of actual physical obstruction. Without validated clinical tools, the current treatment of these symptoms relies primarily on the patient's subjective feedback and the doctor's personal training and experience, which can lead to inconsistent and unsatisfactory outcomes.

Through a series of preliminary studies, the investigators demonstrated that the symptom of nasal obstruction may be caused not by obstruction per se but by poor sensing of airflow during breathing or sensing may be worsened by impaired trigeminal function. However, which trigeminal sensory regions and what nasal airflow anomalies are most critical in disrupting the sensing of airflow are still unknown. In Aim 2, the investigators will investigate the efficacy of a novel patent-pending "nasal aid" to improve patients' symptoms by modulating nasal airflow and trigeminal sensory feedback and to improve future treatment outcomes based on what the investigators have learned and will continue to learn about the airflow trigeminal perception mechanisms.

The outcomes from this research may potentially validate several novel clinical tools to better identify factors that most affect patients' obstructive symptoms and to relieve symptoms by modulating nasal airflow patterns. The ultimate goal is to assist patients and clinicians in planning effective, well-informed, personalized treatment strategies, potentially saving millions of healthcare dollars annually while improving patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Smell Loss complaints
2. Nasal Obstruction

Exclusion Criteria:

1. Congenital olfactory losses
2. Nasal polyps, blocking the olfactory cleft
3. Significant atrophy
4. Cystic fibrosis
5. Wegeners or any other connective tissue disorder
6. Head trauma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Nasal Obstruction Symptom Evaluation (NOSE) questionnaire | 3 time points: 1-baseline, 2-after the applications of nasal aid (done on the first day of testing), and 3- 8 weeks after surgery.
  A clinically validated 5 item questionnaire to document general nasal obstruction. symptoms severity.
Change in Visual Analog Scale (VAS) of nasal obstruction | 3 time points:1-baseline, 2-after the applications of nasal aid (done on the first day of testing) and 3-8 weeks after surgery.
  A visual analog scale of nasal obstruction (VAS), with ratings from 0 to 10 (0 = completely clear; 10 = completely obstructed).
Change in Empty Nose Syndrome 6-Item Questionnaire (ENS 6 Q) | 3 time points:1-baseline, 2-after the applications of nasal aid (done on the first day of testing) and 3-8 weeks after surgery.
  A validated ENS-specific symptom questionnaire.

SECONDARY OUTCOMES:
Change in Sino-nasal Outcome Test (SNOT-22) | 1-baseline (done on the first day of testing)and 2- 8 weeks after surgery
  A validated questionnaire documenting general nasal sinus symptoms.
Change in nasal resistance | 1-baseline (done on the first day of testing) and 2- 8 weeks after surgery
  Anterior rhinomanometry will be used to measure airflow and pressures during normal breathing.
Change in rhinomanometry | 1-Baseline (done on the first day of testing) and 2- 8 weeks post-surgery
  The narrowest area of the nasal airway measured by an acoustic rhinometry.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Zhao, Ph.D, Principal Investigator — Associate Professor
Locations (1):
- Eye and Ear Institute, 915 Olentangy River Road, ENT, Suite 4000, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Formanek VL, Spector BM, Zappitelli G, Wu Z, Zhao K. Designing novel "Smell-Aids" to improve olfactory function in post COVID-19 era. BMC Med. 2025 Mar 24;23(1):169. doi: 10.1186/s12916-025-03999-y. PMID 40128836